CLINICAL TRIAL: NCT07210203
Title: Additional Effects of Neural Mobilization on Pain, Balance and Quality of Life in Diabetic Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/03
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Neuropathy; Postural Balance; Pain
Keywords: Balance; Diabetic Peripheral Neuropathy; Postural Pain; Quality of life
MeSH Terms: conditions — Diabetic Neuropathies; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural moblization with Balance traning (Experimental): Neural Moblization Includes the following protocol:
  Hot Pack 10 mins TENS 10 mins Upper limb and lower limb sliding techniques . (10 reps) Upper limb lower limb tentioning technique (10 reps) Tibial Nerve sliding,Siatic Nerve Sliding,Median nerve Sliding, (10 reps) Combine sliding plue Tensioning,(10 reps) Balance Traning Include:Sitting to standing (10 reps × 2 sets) Standing unsupported (Hold 30s × 3) Standing to sitting (10 reps × 2 sets) Transfers ( 10 reps) Standing with eyes closed( Hold 10-20s ×3) Standing with feet together (Hold 10-20s × 5) Reaching forward with outstretched arm (10 reps) Retrieving object from floor (8-10 reps) Turning to look behind (10 reps each side) Turning 360 degrees (3 reps each) Placing alternate foot on stool(10 reps each) Standing with one foot in front (Hold 15-30s × 3) Standing on one foot( Hold 15-30s × 3) Repetitions will increase gradually week wise
  Interventions: Procedure: Neural mobilization with Balance training with conventional physical Therapy
- Balance traning (Active Comparator): Hot pack 10 mins TENS 10 mins Sitting to standing (10 reps × 2 sets) Standing unsupported (Hold 30s × 3) Standing to sitting (10 reps × 2 sets) Transfers ( 10 reps) Standing with eyes closed( Hold 10-20s ×3) Standing with feet together (Hold 10-20s × 5) Reaching forward with outstretched arm (10 reps) Retrieving object from floor (8-10 reps) Turning to look behind (10 reps each side) Turning 360 degrees (3 reps each) Placing alternate foot on stool(10 reps each) Standing with one foot in front (Hold 15-30s × 3) Standing on one foot( Hold 15-30s × 3) Repetitions will increase gradually week wise
  Interventions: Procedure: Balance Training only with conventional physical therapy

INTERVENTIONS:
Procedure: Neural mobilization with Balance training with conventional physical Therapy — ( HOT pack 10 mins + TENS 10 mins)
  Neural Moblization Includes the following protocol:
  Hot Pack 10 mins TENS 10 mins Upper limb and lower limb sliding techniques . (10 reps) Upper limb lower limb tentioning technique (10 reps) Tibial Nerve sliding,Siatic Nerve Sliding,Median nerve Sliding, (10 reps) Combine sliding plue Tensioning,(10 reps) Balance Training Sitting to standing (10 reps × 2 sets) Standing unsupported (Hold 30s × 3) Standing to sitting (10 reps × 2 sets) Transfers ( 10 reps) Standing with eyes closed( Hold 10-20s ×3) Standing with feet together (Hold 10-20s × 5) Reaching forward with outstretched arm (10 reps) Retrieving object from floor (8-10 reps) Turning to look behind (10 reps each side) Turning 360 degrees (3 reps each) Placing alternate foot on stool(10 reps each) Standing with one foot in front (Hold 15-30s × 3) Standing on one foot( Hold 15-30s × 3) Repetitions will increase gradually week wise
  Arms: Neural moblization with Balance traning
Procedure: Balance Training only with conventional physical therapy — balance training program combines conventional physical therapy with hot pack (10 min) and TENS (10 min), delivered over 4-6 weeks, 3-4 sessions per week, 30-40 minutes each. Training begins with easier Berg Balance Scale (BBS) tasks and progresses as the patient improves.
  In Weeks 1-2, basic static and supported tasks are practiced, including sit-to-stand, standing unsupported (wide to narrow base), supervised transfers, reaching forward, and standing with eyes closed. Weeks 3-4 focus on dynamic stability with picking objects from the floor, head/torso turns, 360° turns, step-ups, and heel-to-toe stance. Weeks 5-6 progress to advanced functional tasks such as alternating foot placement on a stool, tandem stance, one-leg standing, gentle perturbations, and walking 5-10 m with head turns.
  Arms: Balance traning

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) is a common complication of diabetes, affecting up to 50% of patients and causing pain, numbness, and balance impairments, which increase the risk of falls, ulcers, and reduced quality of life. Current treatments mainly manage symptoms, highlighting the need for adjunctive approaches. This randomized controlled trial will evaluate the additional effects of Neural Mobilization (NM) on pain, balance, and quality of life in DPN. Thirty-two patients with type 2 diabetes and DPN will be recruited at Fauji Foundation Hospital and screened using the Michigan Neuropathy Screening Instrument (MNSI). Participants will be randomized into two groups: (1) NM plus Balance Training with standard care and (2) Balance Training alone, each for six weeks (two 30-minute sessions/week). Pain will be assessed using the Numeric Pain Rating Scale (NPRS), balance using the Berg Balance Scale, and quality of life using the Norfolk QOL-DN questionnaire. Outcome measures will be recorded at baseline and post-intervention. Ethical approval will be obtained from FUMC ERC, and data will be analyzed using SPSS v.22.

DETAILED DESCRIPTION:
Diabetic Peripheral Neuropathy (DPN) is a common and debilitating complication of diabetes, affecting nearly 50% of individuals with the condition during their lifetime. It is characterized by nerve damage that leads to symptoms such as pain, numbness, and balance impairments, significantly impacting patients' daily functioning and overall quality of life. The prevalence of DPN is associated with increased risks of falls, foot ulcers, and other serious complications. Current treatment options often focus on managing symptoms but may fall short in addressing the multifactorial nature of the condition. This highlights the urgent need for effective adjunctive therapies that can improve both physical function and quality of life. This study aims to investigate the additional effects of Neural Mobilization (NM) on pain reduction, balance and quality of life improvement, in Diabetic Peripheral Neuropathy (DPN).A randomized controlled trial will be conducted with participants diagnosed with DPN . This study will be a single-blinded, randomized controlled trial with two groups: the intervention group, which will receive Neural Mobilization and Balance Training in addition to standard care, and the control group, which will receive Balance Training alone. The intervention will last for six weeks, with participants attending two 30-minute sessions per week. A total of 32 individuals with type 2 diabetes mellitus and Peripheral Diabetic Neuropathy will be recruited and randomly assigned to one of the two groups. The Michigan Neuropathy Screening Instrument (MNSI) will be used to screen for neuropathy. Quality of life will be measured using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) questionnaire, and pain will be assessed using the Numeric Pain Rating Scale (NPRS). Balance will be assessed by using berg balance scale. The study will be conducted over a period of 1 year at Fauji Foundation Hospital. Ethical approval will be obtained from FUMC ERC. Recruited participants will be allocated to either group through a convenient sampling method. Outcome measurements will be taken at baseline and again after the 6-week intervention period. Individuals meeting the inclusion criteria will be selected, and written informed consent will be obtained after explaining the study's purpose. Data will be entered and analyzed on SPSS v. 22.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Diagnosed cases of Diabetic Peripheral Neuropathy
* Age 50-75 years.
* Patients having history of type 2 Diabetes for at least 5 years.
* Presence of neuropathic symptoms (pain, numbness, tingling, balance issues).
* Patient having mild to moderate pain according to NPRS

Exclusion Criteria:

* Patients with Neurological Disorders like Stroke, multiple sclerosis, Parkinson's disease.
* Chronic Pain Conditions or Conditions unrelated to DPN (e.g., fibromyalgia, osteoarthritis).
* Foot Ulcers/Infection: Active ulcers or infections on lower limbs.
* Uncontrolled Diabetes
* Severe Balance Impairment Individuals unable to perform basic balance tests (e.g., unable to stand unaided for a few seconds).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Pain in Diabetic Neuropathy | 6 weeks
  Numeric Pain Rating Scale (NPRS): 0-10 scale where 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, and 7-10 = severe pain.
Balance | 6 weeks
  Berg Balance Scale (BBS): A 14-item, 0-56 point test of static and dynamic balance where 41-56 = low fall risk, 21-40 = medium fall risk, and 0-20 = high fall risk, with higher scores reflecting better balance and independence.
Quality of life in Diabetic Neuropathy | 6 weeks
  Norfolk QOL-DN total score ranges from -4 to 136. Lower scores reflect better quality of life / fewer neuropathy symptoms, whereas higher scores indicate poorer quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan